CLINICAL TRIAL: NCT07080476
Title: Effectiveness of Kinesio Taping in Patients With Chronic Breast and/or Truncal Oedema After Breast Cancer Treatment: A Randomized Controlled Trial
Brief Title: Effectiveness of Kinesio Taping in Patients With Chronic Breast and/or Truncal Oedema After Treatment for Breast Cancer.
Acronym: KiTaLymph
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiteit Antwerpen (Other)
Collaborators: University Ghent (Other); Iridium Network (Unknown); AZ Groeninge (Unknown)
Responsible Party: Principal Investigator, Nick Gebruers, Associate Professor, Universiteit Antwerpen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 53270
Record Dates: First submitted 2025-07-14; First posted 2025-07-23 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Breast Edema; Breast Cancer Related Lymphoedema; Breast Cancer Related Lymphedema; Truncal Lymphedema
Keywords: RCT; Decongestive Lymphatic Therapy (DLT); Health-related quality of life (HRQoL); Breast cancer; Kinesio taping; Breast oedema
MeSH Terms: conditions — Breast Cancer Lymphedema; Breast Neoplasms | interventions — Athletic Tape

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (standard treatment) (Active Comparator): Participants receive standard DLT, as described in the intervention section, consisting of two sessions per week over four weeks. Self-care activities are continued between sessions and recorded in a self-care diary.
  Interventions: Other: Decongestive lymphatic therapy; Other: Compression bra (sub-study)
- Intervention group (Experimental): Participants receive standard DLT, as described in the intervention section, delivered two times per week over four weeks. In addition, kinesio tape is applied to the affected area by a trained physiotherapist following a standardized protocol. Participants may continue kinesio tape use independently during the follow-up period. A kinesio tape diary is used to record kinesio tape usage.
  Interventions: Other: Decongestive lymphatic therapy; Other: Kinesio tape; Other: Compression bra (sub-study)

INTERVENTIONS:
Other: Decongestive lymphatic therapy — Decongestive lymphatic therapy (DLT) is the current standard of care for lymphoedema management as recommended by the International Society of Lymphology (ISL). It consists of manual lymphatic drainage (MLD), skin care (education), compression therapy using a properly fitted compression bra, and supervised exercise therapy. Sessions last 45 minutes and are delivered two times per week for a period of four weeks.
  On non-treatment days, participants are encouraged to perform home exercises and document self-care practices in a diary.
  Other Names: DLT; complex decongestive therapy
Other: Kinesio tape — Kinesio tape will be applied by trained physiotherapists twice a week. The kinesio tape remains in place for three consecutive days and is replaced once a week. After six days of continuous use, patients will have one rest day without kinesio tape to allow the skin to recover. This cycle will be repeated for the duration of the intervention period.
  The kinesio tape will be applied using a standardised fan-cut technique to ensure consistent application across all study sites. Tape length will be individually tailored. Each application will consist of three fan-shaped strips:
  1. Breast: Anchored at the ipsilateral axilla and directed vertically over the affected breast.
  2. Ventral anastomosis: Originating from the contralateral axilla and applied horizontally over the chest.
  3. Dorsal anastomosis: Also anchored at the healthy axilla and applied horizontally over the back.
  Patients will be instructed in safe self-application for potential use during follow-up.
  Other Names: kinesiotape; kinesio tapes; kinesio taping; kinesiology taping
  Arms: Intervention group
Other: Compression bra (sub-study) — In a subset of participants, different types of commercially available compression bras are tested for pressure and comfort. Each bra is worn for a period of one week without compromising the outcomes of the primary objective. The pressure exerted by the garment is measured using the PicoPress device on the first day of wear. The wearing comfort is evaluated using an adjusted version of the ICC compression questionnaire after one week of wearing the compression bra.

SUMMARY:
The goal of the KiTaLymph trial is to investigate whether the application of kinesio tape is effective in women with persistent (>6 months) breast and/or truncal oedema after treatment for breast cancer.

The main objectives are to assess whether kinesio taping:

* reduces pain and symptoms,
* decreases swelling,
* improves quality of life (QoL).

This study will compare a control group receiving standard care, decongestive lymphatic therapy (DLT), to an intervention group receiving DLT in combination with kinesio taping, in order to determine whether the addition of kinesio tape yields superior clinical outcomes.

Participants will be randomly allocated to one of the two study arms. Both groups will participate in a 4-week intervention phase, consisting of two treatment sessions per week. This will be followed by a 6-month follow-up period to assess the durability of treatment effects and cost-related outcomes.

A total of approximately 128 participants will be recruited. Outcome assessments will be conducted at baseline, immediately post-intervention (1 month), and at 3 and 6 months following the end of the intervention. These assessments will include standardised patient-reported outcome measures evaluating symptoms, quality of life, and pain, namely, the Breast Edema Questionnaire (BrEQ), the EORTC-QLQ-BR23, the EQ-5D-5L, and a visual analogue scale (VAS), as well as objective physical measurements of oedema using the LymphScanner (expressed as percentage water content, PWC).

In addition to the primary research objective, several sub-studies will be conducted. These will include: (1) a longitudinal analysis of the effects of standard treatment; (2) an evaluation of the responsiveness and clinical utility of the BrEQ; and (3) a cross-sectional analysis of the compression pressure exerted by various compression bras. All sub-studies are methodologically feasible within the projected sample size of the primary objective and aim to provide supplementary insights into the clinical management of breast and truncal oedema.

DETAILED DESCRIPTION:
As outlined in the brief summary, three sub-studies will be embedded within the main study sample. The following section provides a concise overview of the methodological approach for each of these sub-studies.

1. The longitudinal effect of decongestive lymphatic therapy:

   This sub-study examines the (long-term) effect of DLT on symptoms and functioning in women with persistent breast and/or truncal oedema following breast cancer treatment. The analysis will focus on participants in the control group, who receive DLT alone. Outcomes such as symptom burden (BrEQ), local tissue water (PWC), pain (VAS), and quality of life (EQ-5D-5L and EORTC-QLQ-BR23) will be tracked at multiple time points: baseline, after 1 month of intervention, and 3 and 6 months after the end of the intervention.

   No additional intervention is introduced beyond the standard treatment already described in the main study protocol. The sub-study will assess the sustainability of symptom improvement over time and provide insight into the standalone effectiveness of DLT.
2. Responsiveness of the Breast Edema Questionnaire:

   This sub-study aims to evaluate the responsiveness of the BrEQ, a validated questionnaire used to assess symptoms related to breast oedema. Although the BrEQ has demonstrated strong psychometric properties, its ability to detect clinically meaningful changes over time has not yet been investigated.

   Participants from both groups in the main study can participate in this sub-study. The design follows a longitudinal cohort structure integrated into the RCT, without any additional interventions. Two subgroups will be analysed: (1) the intensive phase group (from baseline to one month after the start of the intervention), in which clinical improvement is expected, and (2) the maintenance phase group (from three to four months after the end of the intervention), in which symptom levels are expected to remain stable.

   In both groups, BrEQ scores will be compared with patient-reported change using the Global Perceived Effect (GPE) scale. Responsiveness will be quantified through Receiver Operating Characteristic (ROC) curve analysis, and effect size calculations (Cohen's d, standardized response mean). This sub-study requires no additional interventions and uses existing follow-up time points supplemented by one extra BrEQ and GPE assessment at four months after the end of the intervention.
3. Pressure and comfort of compression bras:

This sub-study investigates the pressure exerted by different commercially available compression bras and evaluates patient-reported comfort. The goal is to assess whether these garments provide adequate therapeutic compression and are acceptable for daily use.

The design follows a cross-sectional approach conducted in a subset of participants (five participants per cup size) who consent to this additional component. Each participating patient will receive different compression bras, worn for one week each.

Pressure beneath the garment will be measured using the PicoPress device (Microlab, Italy) on the first day of wear. After each one-week wear period, participants will complete an adapted version of the ICC Compression Questionnaire (ICC-CQ) to assess comfort and usability.

ELIGIBILITY:
Inclusion Criteria:

* Female patients previously treated for breast cancer.
* Suffering from persistent (>6 months) breast and/or truncal oedema, established at least six months after completion of radiotherapy.
* Objective measurements:

  * BrEQ score ≥9.
  * PWC (LymphScanner) showing at least one of the following:

    * Truncal oedema: ratio ≥ 1.32.
    * Breast oedema: ratio ≥ 1.28.
    * Local PWC of 52.90%.
* Clinical evaluation:

  * At least one positive sign of breast and/or truncal oedema such as:

    * Visual swelling compared with the contralateral side.
    * Visible imprint of the bra on the skin.
    * Peau d'orange appearance on the breast.

Exclusion Criteria:

* Presence of skin infections or wounds of the breast/truncal region at the time of inclusion making it impossible to apply kinesio tape.
* Age under 18 years.
* Not able to read and understand Dutch language.
* Having received mastectomy.
* Metastatic breast cancer.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change in Breast Edema Questionnaire (BrEQ) score | From baseline to the end of one month of treatment
  The Breast Edema Questionnaire (BrEQ) is a validated Dutch patient-reported outcome measure designed to assess the impact of breast oedema. Part 1 of the BrEQ evaluates eight symptoms: pain, heaviness, swelling, tensed skin, redness, pitting sign, enlarged skin pores, and hardness. Each symptom is scored on an 11-point Likert scale ranging from 0 ("not at all") to 10 ("very severe"), resulting in a total symptom score ranging from 0 to 80. Higher scores indicate greater severity of breast oedema symptoms. A total score of ≥9 has been identified as the optimal cut-off point to discriminate between patients with and without breast oedema. The primary comparison will assess group differences in BrEQ score after one month of treatment.

SECONDARY OUTCOMES:
Change in local tissue water (PWC) | From baseline to the end of the treatment period (1 month), and 3 and 6 months after the end of the treatment.
  The LymphScanner is a non-invasive diagnostic device used to objectively measure percentage water content (PWC) in subcutaneous tissue. It uses tissue dielectric constant (TDC) technology to assess local water levels. Measurements are taken at standardised points on the breast and trunk from which ratios are calculated to monitor evolution. Higher PWC values indicate higher levels of local tissue water. Changes over time reflect progression or reduction of oedema.
Change in pain intensity (VAS). | From baseline to the end of the treatment period (1 month), and 3 and 6 months after the end of the treatment.
  Pain intensity is assessed with the Visual Analogue Scale (VAS), a validated 10-cm horizontal scale on which participants indicate their perceived pain level. The scores range from 0 (no pain) to 10 (worst pain). The outcome is the change in VAS scores over time. A decrease in score indicates a reduction in pain severity.
Change in quality of life (EORTC-QLQ-BR23). | From baseline to the end of the treatment period (1 month), and 3 and 6 months after the end of the treatment.
  The EORTC-QLQ-BR23 is a breast cancer-specific quality of life questionnaire developed by the European Organisation for Research and Treatment of Cancer (EORTC). It assesses the quality of life in breast cancer patients, focusing on aspects like body image, sexual functioning, treatment side-effects and emotional well-being. Scores for each domain are linearly transformed to a 0-100 scale. Higher scores on functional scales indicate better functioning, while higher scores on symptom scales indicate more severe symptoms.
Change in quality of life (EQ-5D-5L) | From baseline to the end of the treatment period (1 month), and 3 and 6 months after the end of the treatment.
  The EQ-5D-5L is a standardised tool for measuring health-related quality of life in breast cancer patients. It consists of five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each rated on five levels of severity. The questionnaire also includes a visual analogue scale, where patients rate their overall health on a scale from 0 (worst health imaginable) to 100 (best health imaginable). The outcome is the change from baseline in both the index-based utility score and VAS score.
Documentation of self-reported standard care practices using a self-care diary during the intervention and follow-up periods. | From enrollment to the end of the study at 7 months.
  A self-developed diary for standard care, which is a comprehensive tool designed to track various aspects of standard care during the intervention period and follow-up. Its primary purpose is to provide a detailed record of essential care practices, ensuring participants follow the recommended protocols and enabling investigators to monitor progress accurately.
  The diary will cover several key areas: skin care, compression therapy, exercises, physiotherapy and a few additional questions.
Feasibility and self-reported use of kinesio tape during follow-up as documented in a diary (intervention group only). | From the end of the 4-week intervention period to the 6-month follow-up measurement.
  A self-developed diary for assessing the feasibility of kinesio tape application. This diary tracks when the tape is applied, how long it is worn, and evaluates how feasible it is for the patient to apply it independently. Additionally, it monitors costs to determine the cost-effectiveness of kinesio taping.
Change in Breast Edema Questionnaire (BrEQ) score at 3 and 6 months post end of treatment. | From the end of the 4-week intervention period to the 6-months follow-up measurements.
  The BrEQ is a validated patient-reported measure of breast oedema symptoms. Part 1 includes 8 items scored from 0 (not at all) to 10 (very severe), with a total score ranging from 0 to 80. Higher scores indicate worse symptoms. A score of ≥9 indicates presence of breast oedema.
Responsiveness of the BrEQ (substudy) | From baseline to one month of intervention (intensive group); and 3 and 4 months post-intervention (maintenance group).
  The responsiveness of the BrEQ analysed via comparison with the Global Perceived Effect (GPE) scale and ROC analysis. Additional analyses include Cohen's d and SRM.
Pressure under compression bras (substudy) | First day of wearing the compression bra.
  Pressure (in mmHg) exerted by different commercially available compression bras will be measured using the PicoPress device.
Comfort of a compression bra (substudy) | After one week of wearing the specific compression bra.
  Patient-reported comfort is assessed using an adjusted version of the International Compression Club Compression Questionnaire (ICC-CQ), patient version. The questionnaire includes items about putting on and taking off the compression garment, perceived comfort, and any side effects experienced. It consists of yes/no questions and items rated on an 11-point Likert scale (0-10).
  Higher scores indicate greater ease in putting on and taking off the garment, greater comfort, and more side effects, respectively. No total or summary scores are calculated.

CONTACTS AND LOCATIONS:
Locations (4):
- Belgium (4):
  - University of Antwerp, Antwerp
  - Iridium Network, Antwerp
  - Ghent University Hospital, Ghent
  - AZ Groeninge, Kortrijk

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared "as open as possible, as closed as needed", according to the FAIR principles. Data will be made available upon reasonable request.

REFERENCES:
- [Background] Mayrovitz HN, Somarriba C, Weingrad DN. Breast Tissue Dielectric Constant as a Potential Breast Edema Assessment Parameter. Lymphat Res Biol. 2022 Feb;20(1):33-38. doi: 10.1089/lrb.2020.0137. Epub 2021 Mar 24. PMID 33761280
- [Background] Mayrovitz HN, Weingrad DN. Tissue dielectric constant ratios as a method to characterize truncal lymphedema. Lymphology. 2018;51(3):125-131. PMID 30422435
- [Background] Executive Committee of the International Society of Lymphology. The diagnosis and treatment of peripheral lymphedema: 2020 Consensus Document of the International Society of Lymphology. Lymphology. 2020;53(1):3-19. PMID 32521126
- [Background] Mazor M, Smoot BJ, Mastick J, Mausisa G, Paul SM, Kober KM, Elboim C, Singh K, Conley YP, Mickevicius G, Field J, Hutchison H, Miaskowski C. Assessment of local tissue water in the arms and trunk of breast cancer survivors with and without upper extremity lymphoedema. Clin Physiol Funct Imaging. 2019 Jan;39(1):57-64. doi: 10.1111/cpf.12541. Epub 2018 Sep 12. PMID 30207039
- [Background] Verbelen H, Gebruers N, Beyers T, De Monie AC, Tjalma W. Breast edema in breast cancer patients following breast-conserving surgery and radiotherapy: a systematic review. Breast Cancer Res Treat. 2014 Oct;147(3):463-71. doi: 10.1007/s10549-014-3110-8. Epub 2014 Aug 28. PMID 25164973
- [Background] Verbelen H, Tjalma W, Dombrecht D, Gebruers N. Breast edema, from diagnosis to treatment: state of the art. Arch Physiother. 2021 Mar 29;11(1):8. doi: 10.1186/s40945-021-00103-4. PMID 33775252